CLINICAL TRIAL: NCT02956798
Title: Phase II Trial of SAbR for Patients With Oligometastatic Renal Cell Carcinoma
Brief Title: SAbR For Oligometastatic Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042016-046
Record Dates: First submitted 2016-10-26; First posted 2016-11-07 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Oligometastatic Renal Cell Carcinoma
Keywords: Renal Cell, Stereotactic ablative body radiotherapy (SAbR), Pazopanib, Oligo-mets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Stereotactic ablative body radiation (SABR) (Experimental): Stereotactic ablative body radiation (SAbR) to all sites of measurable metastases (≤3) will be treated by SAbR. New sites of metastasis will be evaluated for continued treatment if deemed appropriate by both medical and radiation oncologists with SAbR.
  Interventions: Radiation: Stereotactic ablative body radiation (SABR)

INTERVENTIONS:
Radiation: Stereotactic ablative body radiation (SABR) — SAbR treatment regimens including ≥25Gy x1 fraction, ≥12Gy x 3 fractions, or ≥8Gy x 5 fractions.

SUMMARY:
Hypothesis:

Stereotactic ablative body radiation (SAbR) prolongs progression-free survival for patients with oligometastatic kidney cancer (RCC) and delays the initiation of systemic therapy.

Primary Objectives:

• To evaluate the delay in time to start of systemic therapy (TTST) as a surrogate of progression free survival (PFS), defined as the time from the first day of SAbR to start of systemic therapy.

Secondary Objective:

* To evaluate the modified progression-free survival (mPFS) for patients with oligometastatic renal cell carcinoma who are treated with SAbR.
* To evaluate the overall survival (OS)
* To evaluate the cancer specific survival (CSS)
* To evaluate the local control rate of irradiated lesions.
* To measure the health-related quality of life (HRQOL).

DETAILED DESCRIPTION:
The study is a prospective single institution phase II single-arm open-label trial evaluating SAbR in patients with newly diagnosed oligometastatic RCC.

Problem Statements:

* Can local therapy (SAbR) safely delay the start of systemic therapy?
* Safely delaying the start of systemic therapy can have significant quality of life benefits for patients since systemic therapy has significant side effects.
* Can SAbR be curative in truly oligometastatic RCC patients?

Primary Endpoint:

• Time to start of systemic therapy (TTST) defined as the time from the first day of SAbR to start of systemic therapy.

Secondary Endpoint:

* Modified progression-free survival (mPFS) is defined as the survival interval without development of >3 sites of new metastasis, new sites of metastases that are not amenable to SAbR treatment, a total of >6 sites of metastasis that required SAbR, local failure at SAbR-treated site, or development of brain metastasis.
* Overall Survival
* Local control
* Toxicity
* HRQOL

Sample Size: 23 Patients will be enrolled.

Statistical Analysis: Time to event will be estimated using the Kaplan-Meier approach along with the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell carcinoma with limited measurable extracranial metastases (Limited metastases, or oligometastases, defined as ≤3 sites of metastasis).
* Radiographic evidence of metastatic disease. CT should be performed within 30 days of registration.
* Pathology confirmation of Renal cell carcinoma.
* Prior surgery, or radiation is permitted.
* Age ≥ 18 years.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and for 90 days after Radiation treatment has been completed . Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  * Ability to understand and the willingness to sign a written informed consent and agrees to undergo image studies and follow up

Exclusion Criteria:

* Subjects with brain metastasis as assessed by contrast MRI or contrast CT scans(contrast recommended).
* Subjects with previous history of brain metastasis.
* Subjects that received prior systemic therapy for kidney cancer in the past 1 year, except one line of immuno- or cytokine therapy (e.g. prior IL-2); systemic therapy for other cancers does not apply to this exclusion criteria
* Subjects with ≥3 unfavorable prognostic factors defined by Motzer et al. (1999), (KPS <80% or ECOG>1, Hgb < LLN, LDH >1.5x normal, corrected serum calcium >10mg/dl and absence of prior nephrectomy), Patients with 0, 1-2, and ≥3 factors had time to death of 20 months, 10 months and 4 months.
* Subjects with life expectancy < 6 months.
* Subjects receiving any other investigational agents
* Subjects must not be pregnant due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to start of systemic therapy (TTST) | 1 Year
  To evaluate the delay in time to start of systemic therapy (TTST) as a surrogate of progression free survival (PFS), defined as the time from the first day of SAbR to start of systemic therapy.

SECONDARY OUTCOMES:
Modified progression-free survival (mPFS) for patients who are treated with SAbR | 6 years
  Modified progression-free survival (mPFS) for patients with oligometastatic renal cell carcinoma who are treated with SAbR. Modified progression-free survival (mPFS) is defined as the survival interval without development of >3 sites of new metastasis, new sites of metastases that are not amenable to SAbR treatment, a total of >6 sites of metastasis that required SAbR, local failure at SAbR-treated site, or development of brain metastasis, with the definition of new metastasis and local failure (progression) as defined by RECIST. "Metastasis" in this entire protocol refers to extra-cranial metastasis unless otherwise specified.
Progression-free survival on systemic therapy (mPFS) | 6 years
  To evaluate progression on next line of systemic therapy as defined by RECIST 1.1 starting from mPFS (modified progression free survival). Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1) Committee [Eur J Cancer. 2009;45(2):228-247]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST v1.1 criteria.
Overall survival (OS) | 6 years
  Overall survival (OS), which is defined as the time between date of registration and the date of death due to any cause.
Cancer specific survival (CSS) | 6 years
  Cancer specific survival is defined as the time between date of registration and the date of death due to renal cell carcinoma.
Local Control | 6 years
  Radiographic progression with >30% increase in the longest diameter of the treated lesions.
Median response duration | 6 years
  Median response duration is defined as the time between the date a response (CR or PR) was first seen until date of progression. Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1) Committee [Eur J Cancer. 2009;45(2):228-247]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST v1.1 criteria.
Time to development of new lesions | 6 years
  Interval time to development of new lesions that can be treated with additional local therapy- title would be this or a shortened version of it. Time to event will be estimated using the Kaplan-Meier approach along with the 95% confidence interval.
Time to disease progression that cannot be treated | 6 years
  To measure the time interval from registration to time to disease progression that cannot be treated with further local therapy and need to initiate or switch systemic therapy. Time to event will be estimated using the Kaplan-Meier approach along with the 95% confidence interval.
Acute & Delayed Toxicity | 6 years
  Severity or Toxicity will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0. Dose adjustments should be made according to the system showing the greatest degree of toxicity. The consequences of toxicity should all be graded 1-5 according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 occurring prior to 270 days from the start of protocol treatment. Other treatment related toxicity attributed to the therapy will be captured, recorded and the consequences of should all be graded 1-5 according to the Common Terminology Criteria for Adverse Events (CTCAE). CTCAE V5.0 along with grades 1-5.
Health-related quality of life (HRQOL) FACT-G | 6 years
  HRQOL will be measured using FACT-G questionnaire at baseline and at first follow up 8-12 weeks (+/- 4 weeks) then 12 week (±4 week) intervals for 1 year, and every 26 weeks (±4 weeks) until the completion of follow ups. FACT-G is a measure that sums the functional well being (FWB), physical well being (PWB), the social/family well-being (S/FWB), and emotional well being (EMB).
Health-related quality of life (HRQOL) EQ-5D | 6 years
  HRQOL will be measured using EQ-5D (EuroQol- 5 Dimension) questionnaire at baseline and at first follow up 8-12 weeks (+/- 4 weeks) then 12 week (±4 week) intervals for 1 year, and every 26 weeks (±4 weeks) until the completion of follow ups. EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Health-related quality of life (HRQOL) FKSI | 6 years
  HRQOL will be measured using FKSI questionnaire at baseline and at first follow up 8-12 weeks (+/- 4 weeks) then 12 week (±4 week) intervals for 1 year, and every 26 weeks (±4 weeks) until the completion of follow ups. FKSI adds to the FACT-G (27 items) by including 15 items specific to kidney cancer patients. In a HRQOL study focused on patient with mRCC, a symptoms subscale questionnaire was developed and will also be administered in this study.
Health-related quality of life (HRQOL) cost-effectiveness | 6 years
  Health care utilization data needed to assess costs will be obtained from the cost & convenience questionnaire, which includes costs of hospitalization, treatment, ER visits, physician and clinic visits and medications. Markov modeling with probabilistic sensitivity analysis will be used to correlate quality-adjusted survival and cost. Cost-effective analysis (cost & convenience questionnaire) will be given prior to treatment and at the time of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No